CLINICAL TRIAL: NCT02077972
Title: Whole Body Hyperthermia & Combat-Related Posttraumatic Stress Disorder (PTSD)
Acronym: PTSD + WBH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator transferred to the University of Wisconsin - Madison
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Charles (Chuck) Raison, Clinical Research Professor of Psychiatry, University of Arizona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1216-7558
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Post Traumatic Stress Disorder (PTSD)
Keywords: PTSD; Military service; depression; Whole Body Hyperthermia (WBH)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- High intensity whole-body infrared heating (Experimental): The participant will undergo the WBH intervention where subjects will be induced to levels of heat that increases core body temperature to approximately 37.5-38.5 °C.temperature.
  Interventions: Device: High intensity whole-body infrared heating

INTERVENTIONS:
Device: High intensity whole-body infrared heating — The Whole Body Hyperthermia system uses water-filtered infrared-A (wIRA) heat radiation. The rise in the body's core temperature is correspondingly rapid and well-tolerated. There are two phases of the thermal challenge, 1) Irradiation phase during which the patient lies recumbent with his/her head positioned outside the tent. The wIRA irradiators are arranged above the exposed upper part of the body; and 2) heat retention phase during which the patient lies in the chamber with the walls of the tent positioned to retain heat. Core body temperatures will be raised to those comparable to a mild fever 37.8-38.5°C.

SUMMARY:
Combat-related post traumatic stress disorder (PTSD) has become an increasingly pressing public health problem in the United States following the overseas wars of the last decade. Rates of PTSD have skyrocketed in the military and among veterans, leading to increased rates of suicide, impairment on the job and off, and behavioral changes that negatively affect not just the veteran, but also his or her family. Although effective medication and psychotherapy treatments exist for combat-related PTSD, many individuals suffering with PTSD do not adequately respond to currently available treatment options, highlighting the need to develop and test new interventions for the disorder. To address this pressing clinical issue, the investigators will conduct a pilot study to determine if Whole Body Hyperthermia (WBH) reduces symptoms in adults suffering from combat-related PTSD. The investigators plan to recruit a sample of 10 medically healthy individuals with combat-related PTSD who will receive a single session of WBH to determine if this single session improves PTSD symptoms and, if so, whether this improvement will last at least 2 weeks. To do this, the study will include basic clinical and psychiatric assessments immediately before and one and four weeks after WBH. Because sleep is so often impaired in PTSD, the investigators will measure at-home sleep patterns for a week prior to and a week following the WBH session using sleep diaries and a wristwatch actigraphy device. Given scientific evidence from our research group that WBH may improve depression, the investigators anticipate that it may also be of benefit or adults suffering from combat-related PTSD.

DETAILED DESCRIPTION:
The investigators will direct a clinical trial of Whole Body Hyperthermia (WBH) for treatment of PTSD related to combat exposure. Although the investigators have not yet studied WBH for PTSD, the investigators have data indicating that WBH is effective for the acute treatment of major depression (MDD). Given the high overlap of symptoms between PTSD and Major Depressive Disorder (MDD), as well as the fact that most people with PTSD also meet criteria for MDD, the investigators have reasons for expecting that WBH may also be of benefit for PTSD. The primary objective of the proposed study is to determine if WBH produces improvement in core PTSD symptoms, just as it appears to do in MDD. Indeed, in preliminary studies, a single exposure to WBH resulted in a downward shift in body temperature and a decrease in depressive symptoms as measured using the Center for Epidemiologic Studies Depression Scale (known as the ADS in Germany where this study was conducted) 5 days later. In addition, following exclusion of one patient with bronchopulmonary inflammation that did not show a decrease in body temperature following treatment, a correlation between the shift in body temperature and ΔADS approached statistical significance. These preliminary data are consistent with previous studies showing that 1) patients with seasonal affective disorder in winter during depression have blunted thermoregulatory cooling but have thermoregulatory cooling that is similar in efficiency to control subjects after successful antidepressant response to phototherapy (the retina has direct projections to DRVL serotonergic neurons), 2) ECT increases the circadian amplitude of core body temperature, and decreases mean core body temperature, particularly during the nighttime thermoregulatory cooling period, and 3) thermoregulatory cooling, as evidenced by the number of active sweat glands in depressed patients, increases upon clinical recovery, but not earlier, following ECT. the investigators hypothesize that these relationships in preliminary data and in previous studies are due to dysfunction of the afferent signaling arm of the thermoregulatory system in MDD, specifically the warm afferent system projecting to the LPB and, secondarily, to the DRVL/VLPAG and DRI subsets of serotonergic neurons that have been implicated in anxiolytic and antidepressant actions, respectively, and to normalization of warm afferent signaling following treatment. Again, given the high degree of overlap between PTSD and MDD, the investigators expect that WBH may confer therapeutic benefits in PTSD as it appears to do in MDD.

This clinical trial will only include individuals with PTSD (i.e. no normal controls) in order to determine whether there is a significant effect of a single treatment with WBH administered in an open manner on PTSD symptoms. Based on our data from patients with MDD, the investigators expect that if WBH has an effect on PTSD symptoms, this will be apparent immediately after the treatment and will persist for at least a week. Therefore, the investigators will assess PTSD symptoms prior to and a week following a single treatment with WBH.

Useful preliminary results were obtained from a pilot study comparing mildly to severely depressed patients receiving hyperthermic treatment (N=11) to depressed patients receiving psychotherapy as usual (N=3). Baseline scores on the German language ADS depression scale were similar for the two groups (mean=30.64, sd=9.18, N=11, vs. mean =32.33, sd=17.04, N=3). Raw change on the ADS was significantly greater for the hyperthermia group (mean=-11.91, sd=6.55, N=11, vs. mean=-1.33, sd=4.51, N=3; t=2.60, df=12, P=0.023), resulting in a very large standardized treatment difference (Cohen d) of 1.69 (95% CI=1.00 - 2.48). Percent change was also significant (mean=-39.4, sd=18.9, N=11, vs. mean=-8.6, sd=17.0, N=3; t=2.54; df=12, P=0.026), for a Cohen d of 1.66 (95% CI=0.93 - 2.39). The percentage of the hyperthermia vs. psychotherapy group achieving a clinical response (>50% reduction from baseline) was 27.3% vs. 0%, and the percentage achieving at least a partial response (>25% improvement) was 81.8% vs. 33.3%. These data suggest that our proposed sample size of 10 individuals with combat-related PTSD should be sufficient to identify a potential therapeutic effect, assuming that such an effect would be of similar magnitude to the effect seen in MDD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients aged 18-65.
* Able to understand the nature of the study and able to provide written informed consent prior to conduct of any study procedures.
* A diagnosis of combat-related PTSD based on a PTSD Checklist (PCL)-Military Version score of 50 or greater and meets a diagnosis of PTSD by DSM-V criteria.
* In the investigator's opinion, has met DSM-V criteria for PTSD for at least 4 weeks prior to signing consent.
* Able to communicate in English with study personnel.
* Women of child-bearing potential (i.e., one who is biologically capable of becoming pregnant) must be willing to use a medically acceptable form of birth control or practice abstinence for the duration of her participation in the trial per self-report.

Exclusion Criteria:

* Any of the following diagnoses, as identified by the psychiatric evaluation or study assessments:
* A current DSM-IV-TR Axis I diagnosis of Dementia; or
* Any current DSM-IV-TR Axis II diagnosis (i.e. personality disorder) that would suggest potential noncompliance with the protocol; or
* A lifetime history of Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder Type 1; or
* A diagnosis claustrophobia severe enough that it would impair ability to be in the Heckel HT3000 hyperthermia device
* A current (or within 12 months prior to the Screening visit) diagnosis of Anorexia Nervosa or Bulimia Nervosa
* Subject has met DSM-IV criteria for Substance Abuse in the month prior to screening visit, or non-remitted Substance Dependence in the 2 weeks prior to screening visit.
* A diagnosis of an anxiety or mood disorder that is considered by the investigator to be of greater source of distress or functional impairment than the patient's PTSD diagnosis. Subjects with co-morbid anxiety and mood disorders not excluded above and considered to be of secondary importance will be permitted in the study.
* Participation in concurrent formal psychotherapy during the trial, or in the 2 weeks prior to the screening visit.
* Subject has a medical condition or disorder that is unstable and clinically significant, or could interfere with the accurate assessment of safety or efficacy of treatment, including:
* individuals who are using prescription drugs that may impair thermoregulatory cooling, including diuretics, barbiturates, and beta-blockers, or antihistamines,
* individuals with cardiovascular conditions or problems (uncontrolled hypertension, congestive heart failure, or documented evidence of coronary artery disease)
* individuals with chronic conditions/diseases associated with a reduced ability initiate thermoregulatory cooling, including Parkinson's, multiple sclerosis, central nervous system tumors, and diabetes with neuropathy,
* hemophiliacs/individuals prone to bleeding,
* individuals with a fever the day of study intervention (if so, they will be rescheduled),
* individuals with hypersensitivity to heat,
* individuals with recent acute joint injury (i.e. arthritis),
* individuals with enclosed infections, be they dental, in joints, or in any other tissues,
* Clinically significant, in the investigator's opinion, abnormal findings on screening laboratory tests or physical exam.
* Presence of clinically significant suicide risk, based on the investigator's opinion, or a Columbia Suicide Severity Risk Scale (C-SSRS) suicidal ideation score of 4 or 5. Any suicide attempt within 3 months of the Screening visit is exclusionary.
* Use of any psychotropic medications for 2 weeks (8 weeks for fluoxetine) prior to initiation of the study, with the exception of a stable dosage of benzodiazepine or non-benzodiazepine hypnotic medications (e.g. zolpidem (Ambien), zaleplon (Sonata), eszopiclone (Lunesta), lorazepam (Ativan), diazepam (Valium), clonazepam (Klonopin), alprazolam (Xanax),
* Need for any non-protocol psychotropic medication once enrolled, with the exception of benzodiazepine or non-benzodiazepine hypnotics used at a stable dosage.
* Use of any psychoactive dietary or herbal products in the 2 weeks prior to screening visit 2, or at any time during the trial.
* Women who are pregnant (HCG pregnancy test at screening) or lactating, or who plan to become pregnant during the study.
* Current participation in any clinical trial that might impact results of this one, which includes participation in another clinical trial for depression, as well as drug trials with agents that might affect mood or regulation of body temperature.
* Reasonable likelihood for non-compliance with the protocol for any other reason, in the opinion of the Investigator, prohibits enrollment of subject into the study.
* Obesity and overall size of subject. It will be at the PI's discretion to consider BMI, waist circumference, and body fat composition when determining eligibility and safety of the individual.
* History of peripheral circulatory disease, for example peripheral vascular disease, deep vein thrombosis (DVT), or lymphedema.
* History of a cerebral vascular accident.
* History of stroke, epilepsy or cerebral aneurisms.
* Cancer in the last five years, except for fully resected non-melanoma skin cancer.
* Diabetes mellitus types I or II.
* Any clinically significant autoimmune disease (compensated hypothyroidism allowed).
* Active alcohol/drug abuse in 2 weeks prior to screening for those who have been dependent or have abused on drugs/alcohol in the last 2 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Clinician Assessment of PTSD Scale (CAPS) | Baseline, 1 and 4 weeks post Intervention
  Change in scores between baseline and subsequent assessments will be assessed to determine the effect of WBH on PTSD symptoms.

SECONDARY OUTCOMES:
Change in depression scores over time [Inventory of Depressive Symptomatology-Self Report (IDS-SR)] | Baseline, 1 and 4 weeks following WBH intervention
  Percent change in scores between baseline and subsequent assessments will be assessed.
Change in Scores on the Brief COPE Measure | Baseline, 1 and 4 weeks following WBH Intervention
  Percent change in scores between baseline and subsequent assessments will be assessed.
Change in scores on the Post Traumatic Stress Disorder Checklist (Military) | Baseline, 1 and 4 weeks following the WBH intervention
  Percent change in scores between baseline and subsequent assessments will be assessed using the PCL-Military checklist.
Change in scores on the Primary Care PTSD Screen | Baseline, 1 and 4 weeks following the WBH intervention
  Percent change in scores between baseline and subsequent assessments will be assessed using the Primary Care PTSD Screen.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Raison, MD, Principal Investigator — University of Arizona, Department of Psychiatry, College of Medicine
Locations (1):
- University of Arizona, Tucson, Arizona, United States